CLINICAL TRIAL: NCT04235231
Title: The Effect of Lateral Tilt on Ventilation Distribution in Lungs Assessed by Electrical Impedance Tomography: A Pilot Prospective Randomized Study in Neurocritical Care
Brief Title: The Effect of Lateral Tilt on Ventilation Distribution in Lungs Assessed by Electrical Impedance Tomography
Acronym: N-LAT-EIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital Liberec (Other)
Collaborators: Charles University, Czech Republic (Other); University of Sao Paulo (Other); Technology Agency of the Czech Republic (Unknown)
Responsible Party: Principal Investigator, Vera Spatenkova, MD, Ph.D., Head of Neurocenter, Regional Hospital Liberec
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RHL-NICU-2020-01
Record Dates: First submitted 2020-01-09; First posted 2020-01-21 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Lung Collapse
Keywords: Lung Inhomogeneity; Lung Collapse; Atelectasis; Mechanical Ventilation; EIT; Bed tilting; Positioning; Neurocritical Care; Unconsciousness; Acute Brain Disease; Preventive Strategy
MeSH Terms: conditions — Pulmonary Atelectasis; Unconsciousness | interventions — Posture

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Research Randomizer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral tilt bed (Experimental): Bed tilting (15° lateral tilt, original product brand name LINET Eleganza 5)
  Interventions: Device: Bed tilting
- Body positioning (Experimental): Manual positioning of body by nurse.
  Interventions: Other: Body positioning

INTERVENTIONS:
Device: Bed tilting — 15° lateral tilt, original product brand name LINET Eleganza 5
  Arms: Lateral tilt bed
Other: Body positioning — Manual positioning of body by nurse: left side, back, right side, using positioning pillows
  Other Names: Manual positioning of body by nurse
  Arms: Body positioning

SUMMARY:
Prevention of lung inhomogeneity is an essential part of preventive strategy in neurocritical care, reducing the risks of secondary brain damage from hypoxemia, hypo/hypercapnia or pneumonia.

DETAILED DESCRIPTION:
In the monocentric, intervention, prospective, randomized study, the investigators will examine the effect of lateral tilting (routinely used in critical care) on the lung inhomogeneity that will be analyzed by electrical impedance tomography (EIT) in the unconscious patients with acute primary brain disease and artificial pulmonary ventilation. Two types of lateral tilting will be compared: manual positioning of body by nurse versus the bed tilting (15° lateral tilt, original company (LINET) and product brand name (Eleganza 5).

ELIGIBILITY:
Inclusion Criteria:

* Primary brain disease
* Hospitalization in Neurocenter, Neurointensive Care Unit
* Age>18 years
* Unconsciousness
* Artificial pulmonary ventilation

Exclusion Criteria:

* Intracranial hypertension
* History of primary lung disease
* The terminal stage of the disease
* Refractory hemodynamic instability

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Atelectasis/collapse | up to 24 weeks
  Assessed by electrical impedance tomography (EIT) or chest x-ray (CXR) at end of observation period

SECONDARY OUTCOMES:
Evaluating oxygenation parameters | up to 24 weeks
  Oxygen saturation
Evaluating hemodynamic parameters | up to 24 weeks
  Hemodynamic monitoring: stroke volume variation (SVV)
Cost effectiveness measurement between two groups | up to 24 weeks
  Therapeutic Intervention Scoring System (TISS)
Profiling pneumonia incidence | up to 24 weeks
  Pneumonia score
Comparing duration of stay in Neurocenter Neurointensive Care Unit | up to 24 weeks
  Days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Vera Spatenkova, MD, Ph.D., Study Chair — NeuroCenter
Locations (1):
- Regional Hospital Liberec, Liberec, Czechia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT04235231/Prot_SAP_000.pdf